CLINICAL TRIAL: NCT00491036
Title: Randomized Clinical Study of Intraaortic Balloon Pump Use in Cardiogenic Shock Complicating Acute Myocardial Infarction
Brief Title: Intraaortic Balloon Pump in Cardiogenic Shock II
Acronym: IABP-SHOCK II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Holger Thiele, Deputy Director, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 342
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Myocardial Infarction; Shock, Cardiogenic
Keywords: Acute myocardial infarction; cardiogenic shock; percutaneous coronary intervention; intraaortic balloon counterpulsation; Acute myocardial infarction - cardiogenic shock
MeSH Terms: conditions — Myocardial Infarction; Shock, Cardiogenic | interventions — Intra-Aortic Balloon Pumping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intraaortic balloon pump (Active Comparator): Patients in cardiogenic shock get an intraaortic balloon pump in the cath lab
  Interventions: Device: Intraaortic balloon pump
- No intraaortic balloon pump (No Intervention): Patients in cardiogenic shock in this group get no intraaortic balloon pump

INTERVENTIONS:
Device: Intraaortic balloon pump — intraaortic balloon pump from Datascope/Maquet or Arrow/Teleflex will be used
  Arms: Intraaortic balloon pump

SUMMARY:
Patients in cardiogenic shock complicating acute myocardial infarction (AMI) are referred to a tertiary care center for percutaneous coronary intervention (PCI) of the infarct related artery in this multicenter, ran-domized clinical trial. After checking in- and exclusion criteria computerized randomization is performed to either PCI plus intraaortic balloon pump (IABP) insertion and medical treatment or PCI plus medical treatment only. Intensive care treatment is performed according to standard care including hemodynamic monitoring using a pulmonary artery catheter for optimal volume status adaptation and inotropic drug administration.

The IABP will be weaned after hemodynamic stabilization. Primary outcome measure will be 30-day mortality. The secondary outcome measures such as hemody-namic, laboratory and clinical parameters will serve as surrogate for prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

Cardiogenic shock complicating acute myocardial (STEMI or NSTEMI) with

* intended revascularization (PCI or CABG)
* Systolic blood pressure < 90 mmHg > 30 min or inotropes required to maintain pressure > 90 mmHg during systole
* Signs of pulmonary congestion
* Signs of impaired organ perfusion with at least one of the following:

  * Altered mental status
  * Cold, clammy skin
  * Urine output <30 ml/h
  * Serum lactate >2mmol/l
* Informed consent

Exclusion criteria:

* Resuscitation > 30 minutes
* Cerebral deficit with fixed dilated pupils
* No intrinsic heart action
* Mechanical infarction complication
* Onset of shock > 12 h
* Severe peripheral artery disease
* Aortic regurgitation > II.°
* Age > 90 years
* shock of other cause
* Other severe concomitant disease
* participation in another trial

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 day

SECONDARY OUTCOMES:
Inflammatory markers (CRP and white blood cell count) | 4 days
Hemodynamic Parameters (Blood pressure, Heart rate) | 3 days
Time till hemodynamic stabilization | 30 days
Catecholamine dose and duration of catecholamines | 30 days
Mean and area under the curve of serum lactate | 48 hours
Creatinine clearance until stabilization | 4 days
requirement for hemofiltration or dialysis | 4 days
length of ICU stay | 30 days
length of mechanical ventilation | 30 days
SAPS-II Score | 4 days
requirement for active assist device implantation or heart transplantation at 30 days and approximately 60 months | 60 months
long-term mortality at 6, 12 and approximately 60 months | 60 months
quality of life at 30 days and approximately 60 months | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Study Chair — Heart Center Leipzig - University Hospital
Locations (20):
- Germany (20):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Segeberger Kliniken Gmbh, Bad Segeberg
  - Charité Berlin, Campus Benjamin Franklin, Berlin
  - Heart Center Bernau - Brandenburg, Bernau
  - Herzzentrum Cottbus, Cottbus
  - Klinikum Lippe-Detmold, Detmold
  - Krankenhaus Fulda, Fulda
  - University Greifswald, Greifswald
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - SLK-Kliniken Heilbronn, Heilbronn
  - Oberhavel-Kliniken Hennigsdorf, Hennigsdorf
  - Klinikum der Universität Jena, Jena
  - Asklepios Klinik Langen, Langen
  - University of Leipzig - Heart Center, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen
  - University of Lübeck, Lübeck
  - Otto-von-Guericke University Magdeburg, Magdeburg
  - German Heart Center Munich, Munich
  - Krankenhaus der Barmherzigen Brüder, Regensburg

REFERENCES:
- [Derived] Lehrke M, Fuernau G, Jung C, Kahles F, Moellmann J, Eitel I, Thelemann N, Desch S, Werdan K, Zeymer U, Adams V, Marx N, Thiele H. GLP-1 in patients with myocardial infarction complicated by cardiogenic shock-an IABP-SHOCK II-substudy. Clin Res Cardiol. 2024 Aug;113(8):1211-1218. doi: 10.1007/s00392-023-02366-2. Epub 2024 Jan 3. PMID 38170249
- [Derived] Ceglarek U, Schellong P, Rosolowski M, Scholz M, Willenberg A, Kratzsch J, Zeymer U, Fuernau G, de Waha-Thiele S, Buttner P, Jobs A, Freund A, Desch S, Feistritzer HJ, Isermann B, Thiery J, Poss J, Thiele H. The novel cystatin C, lactate, interleukin-6, and N-terminal pro-B-type natriuretic peptide (CLIP)-based mortality risk score in cardiogenic shock after acute myocardial infarction. Eur Heart J. 2021 Jun 21;42(24):2344-2352. doi: 10.1093/eurheartj/ehab110. PMID 33647946
- [Derived] Fuernau G, Desch S, de Waha-Thiele S, Eitel I, Neumann FJ, Hennersdorf M, Felix SB, Fach A, Bohm M, Poss J, Jung C, Ouarrak T, Schneider S, Werdan K, Zeymer U, Thiele H. Arterial Lactate in Cardiogenic Shock: Prognostic Value of Clearance Versus Single Values. JACC Cardiovasc Interv. 2020 Oct 12;13(19):2208-2216. doi: 10.1016/j.jcin.2020.06.037. PMID 33032708
- [Derived] Thiele H, Zeymer U, Thelemann N, Neumann FJ, Hausleiter J, Abdel-Wahab M, Meyer-Saraei R, Fuernau G, Eitel I, Hambrecht R, Bohm M, Werdan K, Felix SB, Hennersdorf M, Schneider S, Ouarrak T, Desch S, de Waha-Thiele S; IABP-SHOCK II Trial (Intraaortic Balloon Pump in Cardiogenic Shock II) Investigators; IABP-SHOCK II Investigators. Intraaortic Balloon Pump in Cardiogenic Shock Complicating Acute Myocardial Infarction: Long-Term 6-Year Outcome of the Randomized IABP-SHOCK II Trial. Circulation. 2019 Jan 15;139(3):395-403. doi: 10.1161/CIRCULATIONAHA.118.038201. Epub 2018 Nov 11. PMID 30586721
- [Derived] Poss J, Koster J, Fuernau G, Eitel I, de Waha S, Ouarrak T, Lassus J, Harjola VP, Zeymer U, Thiele H, Desch S. Risk Stratification for Patients in Cardiogenic Shock After Acute Myocardial Infarction. J Am Coll Cardiol. 2017 Apr 18;69(15):1913-1920. doi: 10.1016/j.jacc.2017.02.027. PMID 28408020
- [Derived] Ledwoch J, Fuernau G, Desch S, Eitel I, Jung C, de Waha S, Poess J, Schneider S, Schuler G, Werdan K, Zeymer U, Thiele H. Drug-eluting stents versus bare-metal stents in acute myocardial infarction with cardiogenic shock. Heart. 2017 Aug;103(15):1177-1184. doi: 10.1136/heartjnl-2016-310403. Epub 2017 Feb 7. PMID 28174212
- [Derived] Jung C, Fuernau G, Eitel I, Desch S, Schuler G, Kelm M, Adams V, Thiele H. Incidence, laboratory detection and prognostic relevance of hypoxic hepatitis in cardiogenic shock. Clin Res Cardiol. 2017 May;106(5):341-349. doi: 10.1007/s00392-016-1060-3. Epub 2016 Dec 8. PMID 27928583
- [Derived] Zeymer U, Werdan K, Schuler G, Zahn R, Neumann FJ, Furnau G, de Waha S, Schneider S, Thiele H. Editor's Choice- Impact of immediate multivessel percutaneous coronary intervention versus culprit lesion intervention on 1-year outcome in patients with acute myocardial infarction complicated by cardiogenic shock: Results of the randomised IABP-SHOCK II trial. Eur Heart J Acute Cardiovasc Care. 2017 Oct;6(7):601-609. doi: 10.1177/2048872616668977. Epub 2016 Sep 21. PMID 27655918
- [Derived] Poss J, Fuernau G, Denks D, Desch S, Eitel I, de Waha S, Link A, Schuler G, Adams V, Bohm M, Thiele H. Angiopoietin-2 in acute myocardial infarction complicated by cardiogenic shock--a biomarker substudy of the IABP-SHOCK II-Trial. Eur J Heart Fail. 2015 Nov;17(11):1152-60. doi: 10.1002/ejhf.342. Epub 2015 Sep 3. PMID 26333723
- [Derived] Jung C, Fuernau G, de Waha S, Eitel I, Desch S, Schuler G, Figulla HR, Thiele H. Intraaortic balloon counterpulsation and microcirculation in cardiogenic shock complicating myocardial infarction: an IABP-SHOCK II substudy. Clin Res Cardiol. 2015 Aug;104(8):679-87. doi: 10.1007/s00392-015-0833-4. Epub 2015 Feb 27. PMID 25720332
- [Derived] Jung C, Fuernau G, Muench P, Desch S, Eitel I, Schuler G, Adams V, Figulla HR, Thiele H. Impairment of the endothelial glycocalyx in cardiogenic shock and its prognostic relevance. Shock. 2015 May;43(5):450-5. doi: 10.1097/SHK.0000000000000329. PMID 25692257
- [Derived] Schuster A, Faulkner M, Zeymer U, Ouarrak T, Eitel I, Desch S, Hasenfuss G, Thiele H. Economic implications of intra-aortic balloon support for myocardial infarction with cardiogenic shock: an analysis from the IABP-SHOCK II-trial. Clin Res Cardiol. 2015 Jul;104(7):566-73. doi: 10.1007/s00392-015-0819-2. Epub 2015 Jan 31. PMID 25637294
- [Derived] Fuernau G, Poss J, Denks D, Desch S, Heine GH, Eitel I, Seiler S, de Waha S, Ewen S, Link A, Schuler G, Adams V, Bohm M, Thiele H. Fibroblast growth factor 23 in acute myocardial infarction complicated by cardiogenic shock: a biomarker substudy of the Intraaortic Balloon Pump in Cardiogenic Shock II (IABP-SHOCK II) trial. Crit Care. 2014 Dec 21;18(6):713. doi: 10.1186/s13054-014-0713-8. PMID 25528363
- [Derived] Fuernau G, Poenisch C, Eitel I, de Waha S, Desch S, Schuler G, Adams V, Werdan K, Zeymer U, Thiele H. Growth-differentiation factor 15 and osteoprotegerin in acute myocardial infarction complicated by cardiogenic shock: a biomarker substudy of the IABP-SHOCK II-trial. Eur J Heart Fail. 2014 Aug;16(8):880-7. doi: 10.1002/ejhf.117. Epub 2014 Jun 5. PMID 24903195
- [Derived] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, de Waha A, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Lauer B, Bohm M, Ebelt H, Schneider S, Werdan K, Schuler G; Intraaortic Balloon Pump in cardiogenic shock II (IABP-SHOCK II) trial investigators. Intra-aortic balloon counterpulsation in acute myocardial infarction complicated by cardiogenic shock (IABP-SHOCK II): final 12 month results of a randomised, open-label trial. Lancet. 2013 Nov 16;382(9905):1638-45. doi: 10.1016/S0140-6736(13)61783-3. Epub 2013 Sep 3. PMID 24011548
- [Derived] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912